CLINICAL TRIAL: NCT06246396
Title: Antihypertensive Mechanisms of Minocycline in Resistant Hypertension: Role of the Gut Microbiota-brain-immune Axis
Brief Title: Antihypertensive Mechanisms of Minocycline in Resistant Hypertension
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Emory University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202301939; 2R01HL132448-05A1 (NIH)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-01

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: minocycline; blood pressure
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minocycline Hydrochloride (Experimental): Minocycline hydrochloride 100 mg, administered twice daily for 3 months
  Interventions: Drug: Minocycline Hydrochloride
- Placebo (Placebo Comparator): Placebo administered twice daily for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline Hydrochloride — Minocycline Hydrochloride 100 mg twice daily
  Other Names: Minocycline; Minocin
  Arms: Minocycline Hydrochloride
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the mechanisms by which minocycline effect blood pressure in individuals with treatment-resistant hypertension. The main questions it aims to answer are:

* To what extent does minocycline lower blood pressure?
* Are such blood pressure effects mediated through changes in gut microbiota, gut leakiness, systemic inflammation, neuroinflammation, or some combination of these?

Participants will be randomly assigned to treatment with minocycline or placebo, treated daily for 3 months, to evaluate these questions.

DETAILED DESCRIPTION:
One hundred twenty patients with treatment-resistant hypertension will be enrolled. A total of 34 patients (17 from each treatment arm), who are participants in the main study, will also be enrolled in a substudy that includes neuroimaging. The study will last 3 months, and will include 3 visit time points (screening, randomization visit, 3-month follow-up visit).

Participants will be randomly assigned, in a 1:1 allocation, to minocycline 100 mg twice per day, or matching placebo, each provided by the study, and investigators will be blinded to treatment assignment.

At the baseline and 3-month follow-up visit, subjects will undergo:

* A comprehensive medical history and examination, including assessment of antihypertensive treatment history
* A series of behavioral activity questionnaires
* Blood tests (plasma renin activity, aldosterone, catecholamines, serum creatinine, lipid panel, hemoglobin a1c, as well as various biomarkers of immune and inflammatory activity, and gut leakiness markers)
* Urine/saliva tests for antihypertensive adherence
* Gut microbiota profiling via whole metagenomic sequencing of stool samples
* Blood pressure (BP) measurement, including unattended office BP and 24-hour ambulatory BP

Subjects enrolled in the neuroimaging substudy will also have PET/MR imaging performed at each visit. Neuroimaging activities will take place at Emory University in Atlanta, GA.

At the final visit (3-month follow-up), participants will also have blood tests to measure study drug concentration, as a measure of adherence to the assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Uncontrolled TRH, defined as uncontrolled blood pressure (mean 24-hour ambulatory systolic BP ≥125 mm Hg or diastolic BP ≥80 mm Hg) while being adherent to a stable (no changes in ≥14 days prior) antihypertensive regimen of 3 or more drugs, including an adequately dosed diuretic or unable to tolerate a diuretic.
* The participant agrees to have all study procedures performed

Exclusion Criteria:

* Known hypersensitivity or contraindication to minocycline or other tetracyclines
* Recent (≤3 months prior), ongoing, or expected use of oral antibiotics
* Estimated glomerular filtration rate (eGFR) of <45mL/min/1.73m2, using the MDRD equation
* Known secondary hypertension
* History of hypertensive crisis, defined as any in-patient hospitalizations for hypertensive crisis/emergency within the past year
* History of orthostatic hypotension, defined as two or more episode(s) of orthostatic hypotension (reduction of SBP of >20 mm Hg or DBP of >10 mm Hg within 3 minutes of standing) in the past year
* History of myocardial infarction, unstable angina, syncope, or cerebrovascular accident in prior 6 months
* Evidence of alcoholism or drug abuse
* Severe comorbid conditions (i.e., neoplasms or HIV positive or AIDS)
* Current pregnancy or anticipated pregnancy during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
24-h systolic blood pressure | 3 months
  Change in mean 24-hour ambulatory systolic blood pressure
Gut microbiome | 3 months
  Change in butyrate-producing gene abundance
Gut inflammation and leakiness | 3 months
  Change in gut-homing inflammatory T-helper cells
Neuroinflammation | 3 months
  Change in [18F]FEPPA radiotracer uptake on PET/MR imaging

SECONDARY OUTCOMES:
Mucin-degrading gene abundance | 3 months
  Change in mucin-degrading gene abundance
IgA+ coated plasma cells | 3 months
  Change in IgA+ coated plasma cells
Gut leakiness markers | 3 months
  Change in gut leakiness markers, including lipocalin-2, intestinal fatty-acid binding protein (I-FABP), zonulin, and lipopolysaccharides (LPS)
24-h diastolic blood pressure | 3 months
  Change in mean 24-hour diastolic blood pressure
24-h heart rate | 3 months
  Change in mean 24-hour heart rate
Adverse Events | 3 months
  Incidence of treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Smith, PharmD, MPH, Principal Investigator — University of Florida
Locations (1):
- UF Clinical Research Center (UF CRC) - CTSI, Gainesville, Florida, United States